CLINICAL TRIAL: NCT01664962
Title: Search for Genetic Basis of Vulvodynia
Status: Completed | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Prof. Jacob Bornstein, Principal Investigator, Western Galilee Hospital-Nahariya
Other Study IDs: 920080002
Record Dates: First submitted 2012-08-09; First posted 2012-08-14 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Vulvodynia
MeSH Terms: conditions — Vulvodynia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Patients: Women with severe Vulvodynia
- Healthy controls: Women without vulvodynia

SUMMARY:
The purpose of this study is to investigate the possibility of an association between Localized Provoked Vulvodynia (LPV) that is both severe and primary and polymorphic markers/single nucleotide polymorphisms (SNPs) in and around the genes encoding heparanase (HSPE-1), Vanilloid Receptor VR1 (TRPV1), and Nerve Growth Factor (NGF).

DETAILED DESCRIPTION:
The short-term goal proposed for the current study was to investigate the possibility of an association between Localized Provoked Vulvodynia (LPV) that is both severe and primary and polymorphic markers/single nucleotide polymorphisms (SNPs) in and around the genes encoding heparanase (HSPE-1), Vanilloid Receptor VR1 (TRPV1), and Nerve Growth Factor (NGF).

Eight polymorphic SNPs in the three different genes suspected to be involved in LPV has been examined as follow:

1. HSPE gene: Four polymorphic SNPs: rs4693608, rs11099592, rs6856901 and rs4364254 that were found to be informative in the Ashkenazi Jewish population
2. TRPV1 gene: Two polymorphic SNPs: rs222747 and rs8065080.
3. NGF gene: A novel T to C SNP in the promoter region at position -198 (rs11102930) and rs6330 which was found to be associated with anxiety-related personality traits and has been suggested to may affect intracellular processing and secretion of NGF.

ELIGIBILITY:
Inclusion Criteria:o meeting Friedrich's criteria [50] for vulva vestibulitis syndrome

* diagnosed by a gynecological examination with LPV
* diagnosed with a severe degree of the syndrome according to Marinoff [48]
* classified with the primary type of the syndrome according to an interview
* with both parents of Ashkenazi origin.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Vulvodynia, Normal healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2008-11; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Genetic association of Vulvodynia | four years
  the possibility of an association between Localized Provoked Vulvodynia (LPV) that is both severe and primary and polymorphic markers/single nucleotide polymorphisms (SNPs) in and around the genes encoding heparanase (HSPE-1), Vanilloid Receptor VR1 (TRPV1), and Nerve Growth Factor (NGF).

CONTACTS AND LOCATIONS:
Locations (1):
- Western Galilee Hospital, Nahariya, Israel